CLINICAL TRIAL: NCT06927505
Title: Comparative Effects of Unstable Surfaces and Bobath Based Trunk Exercises on Trunk Impairment, Postural Control and Balance in Stroke Patients.
Brief Title: Comparative Effects of Unstable Surfaces and Bobath on Trunk Impairment, Posture and Balance in Post Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0261 Qaila Tariq
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Bobath Approach; Stroke; Balance; Posture
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and outcome assessor were blinded in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (bobath based trunk control training) (Experimental): Participants in this arm will perform bobath based trunk control training for 3 days per week.
  Interventions: Other: Bobath based trunk control training
- Group B (unstable surface trunk training) (Experimental): Participants in this arm will perform unstable surface trunk training for 3 days per week.
  Interventions: Other: Unstable surface trunk training

INTERVENTIONS:
Other: Bobath based trunk control training — Participants in the Bobath based trunk training group will undergo a comprehensive intervention encompassing strengthening exercises, stretching exercises, and motor training. This group will experience a 60-minute session, including 40 minutes of Bobath based exercises along with 20 minutes routine physical therapy. 1. Strengthening the oblique abdominals 2. Weight Shifting (Side-to-Side & Forward-Backward) 3. Pelvic Tilts 4. Functional strengthening of trunk extensors 5. Reaching 6. Latissimus dorsi stretching exercise 7. Bridging 8. Trunk rotation (supine and standing position) 9. Sitting to Standing Transitions (with emphasis on trunk control) 10. Standing Weight Shifts There will be a rest of 1 minute between each set of exercise. Progression of exercises with increase in intensity and resistance.
  Arms: Group A (bobath based trunk control training)
Other: Unstable surface trunk training — This group will receive 60-minute training session that consists of 40 minutes of unstable surfaces exercises and 20 minutes of routine physical therapy 3 days per week for a total of 12 weeks.
  Hook-lying position: (1) Abdominal draw-in maneuver with ball under the buttocks.
  (2) Abdominal muscles isometric contraction. (3) Bridging combining with abdominal draw-in maneuver. Each exercise will be performed with 5-8 repetitions. Sitting: (1) Seated balance (2) Weight shifting e.g. anterior, posterior, lateral (3) Pelvic tilts e.g. anterior and posterior tilt (4) Trunk flexion, extension and lateral flexion on both sides (5) trunk rotation on both sides (6) Reaching e.g. lateral, forward and upward reach (7) Marching while seated Each exercise will be performed with 5-8 repetitions.
  Arms: Group B (unstable surface trunk training)

SUMMARY:
Stroke is an acute, focal neurological deficit attributed to vascular injury (infarction, hemorrhage) of the central nervous system. Trunk control, balance and posture are often impaired after stroke. Trunk and lower limb balance are vital for stroke patients as they significantly impact their functional independence, mobility, and safety. Training on unstable surfaces enhances core strength, balance, coordination, and proprioception. Bobath approach emphasizes the use of controlled, functional movements to enhance postural control and stability. This study aims to determine the comparative effectiveness of trunk training on unstable surfaces and bobath approach on trunk impairment, postural control and balance in stroke patients. The sample size will consist of 45 participants. Group A (unstable surfaces trunk training) and Group B (bobath based trunk training) will receive treatment session of 60 minutes for 3 days per week for 12 weeks. Data will be collected using various assessment tools, including the Trunk impairment scale, Berg balance scale and Postural Assessment Scale for Stroke (PASS) in stroke patients. Assessment will be carried out at baseline, 4th week, 8th week, 12th week and at 16th week after discontinuation of treatment. The data will be entered and analyzed using SPSS version 26. Repeated measures ANOVA will be performed for the with-in group analysis, whereas between-group analysis will be performed using one-way ANOVA.

DETAILED DESCRIPTION:
Trunk control and sitting balance are often impaired after stroke. Patients who are able to sit independently in the early stages after a stroke seem to have greater chances of walking independently at discharge. These impairments are characterized by a diminished siting balance, trunk coordination and muscle strength. In contrast to the extremities, the trunk is bilaterally impaired. Therefore, both the paretic and non-paretic side of the trunk are characterized by reduced activity levels, delayed onset times, and diminished synchronization of the trunk musculature. Therefore, knowledge concerning changes in trunk biomechanics after stroke should be increased so that they can be addressed adequately in therapy. Impaired balance and postural control are an important clinical feature after stroke.

So, incorporating exercises aiming to improve trunk control early in a stroke rehabilitation program should be beneficial for regaining activities of daily living. Trunk rehabilitation is an effective strategy for improving trunk control and sitting balance in addition to finding carryover effects on standing balance and mobility. Swiss ball is widely used for recreational & rehabilitation training programs. As the liable surface of the Swiss ball provides greater challenge for the dynamic balance, co-ordination and trunk control. Swiss exercises facilitate postural control, trunk control, sitting & dynamic balance control by reducing impaired balance & co-ordination by maintaining interaction between nervous system, musculoskeletal system & contextual effects. The Bobath Concept is referred to as the neuro-developmental technique (NDT) worldwide. Stroke patients shall actively participate in exercises assisted by the therapist. Therapists use key points of handling and reflex inhibiting patterns for performing exercises. Bobath approach works on the different types of movement dysfunctions and is based on the active involvement of the patients so that they can develop motor control. This type of therapy incorporates improved functional control and independence. NDT/Bobath concept has been recognized as a treatment for stroke patients with movement dysfunctions. Despite numerous studies investigating rehabilitation techniques for post-stroke patients, there is a notable gap in directly comparing the effects of unstable surface and Bobath-based trunk exercises on trunk impairment, postural control, and balance. Literature is also available about the effectiveness of each intervention in isolation, but according to researcher's knowledge, studies on the comparative effect of these two interventions on trunk control, posture and balance and determining the long-term effects of both types of intervention in stroke have not been conducted yet. So, this study aims to compare the effects of unstable surfaces and Bobath approach on trunk coordination, balance and functional enhancement in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling given criteria will be included in this study:

* Subjects with first onset of stroke.
* Minimum duration for onset of stroke is (3-6) months.
* Subjects aged 25 to 65 years.
* Both male and female genders.
* Patients who are able to follow command.
* Patients who are able to sit independently for 30 seconds.
* MoCA (Montreal Cognitive Assessment) of ≥ 26/30 indicating intact Cognition.

Exclusion Criteria:

Participants having given criteria will be excluded from this study:

* Patient with recurrent attacks.
* Patients who are not able to follow command.
* Patients who have severe limitations in passive range of motion at lower extremities.
* Patients undergoing any other balance training protocol.
* Patients with contraindications to exercise, preexisting neurological disorders, severe communication impairments and history of diagnosed musculoskeletal disorders.
* Patients who are unable to sit independently for 30 seconds.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Trunk impairment scale (TIS) | 4th week
  The Trunk Impairment Scale (TIS) is use to evaluate trunk control. It consists of 17 parameters and evaluates static and dynamic sitting balance and trunk coordination. A higher score indicates better performance. Its validity and reliability have been demonstrated in patients with stroke.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 4th week
  BBS is postural balance scale containing 14 items including standing and sitting unsupported, reaching forward, and placing the alternating foot on a stool. Administering the BBS takes approximately 15 min. Each of the 14 items are scored on a 5-level ordinal scale from 0 ("unable to perform or requiring help") to 4 ("normal performance"), thus providing a potential maximum score of 56 points.
Postural Assessment Scale for Stroke (PASS) | 4th week
  PASS is a scale that makes postural evaluation of patients with stroke in three different positions (i.e. lying, sitting, and standing). The scale consists of 12 items. It is a 4-point type scoring ranging from 0 to 3 points. Total scoring varies between 0 and 36. There are two subscales: "maintaining posture" and "changing posture". Both sections can be scored separately and the sum of these scores gives the total score.

OTHER OUTCOMES:
MoCA (Montreal Cognitive Assessment) | 4th week
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Faisal Masood Teaching Hospital, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva PB, Mrachacz-Kersting N, Oliveira AS, Kersting UG. Effect of wobble board training on movement strategies to maintain equilibrium on unstable surfaces. Hum Mov Sci. 2018 Apr;58:231-238. doi: 10.1016/j.humov.2018.02.006. Epub 2018 Mar 12. PMID 29499471
- [Background] Sag S, Buyukavci R, Sahin F, Sag MS, Dogu B, Kuran B. Assessing the validity and reliability of the Turkish version of the Trunk Impairment Scale in stroke patients. North Clin Istanb. 2018 Aug 14;6(2):156-165. doi: 10.14744/nci.2018.01069. eCollection 2019. PMID 31297483
- [Background] Lee PY, Huang JC, Tseng HY, Yang YC, Lin SI. Effects of Trunk Exercise on Unstable Surfaces in Persons with Stroke: A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Dec 7;17(23):9135. doi: 10.3390/ijerph17239135. PMID 33297451
- [Background] Pathak A, Gyanpuri V, Dev P, Dhiman NR. The Bobath Concept (NDT) as rehabilitation in stroke patients: A systematic review. J Family Med Prim Care. 2021 Nov;10(11):3983-3990. doi: 10.4103/jfmpc.jfmpc_528_21. Epub 2021 Nov 29. PMID 35136756
- [Background] Arienti C, Lazzarini SG, Pollock A, Negrini S. Rehabilitation interventions for improving balance following stroke: An overview of systematic reviews. PLoS One. 2019 Jul 19;14(7):e0219781. doi: 10.1371/journal.pone.0219781. eCollection 2019. PMID 31323068
- [Background] Van Criekinge T, Hallemans A, Herssens N, Lafosse C, Claes D, De Hertogh W, Truijen S, Saeys W. SWEAT2 Study: Effectiveness of Trunk Training on Gait and Trunk Kinematics After Stroke: A Randomized Controlled Trial. Phys Ther. 2020 Aug 31;100(9):1568-1581. doi: 10.1093/ptj/pzaa110. PMID 32542356